CLINICAL TRIAL: NCT03156621
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Alirocumab in Patients With Homozygous Familial Hypercholesterolemia
Brief Title: Study in Participants With Homozygous Familial Hypercholesterolemia (HoFH)
Acronym: ODYSSEY HoFH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R727-CL-1628; 2017-000351-95 (EudraCT Number)
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Results first posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Homozygous Familial Hypercholesterolemia
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia | interventions — alirocumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Alirocumab SC Q2W (Experimental): Alirocumab SC every 2 weeks (Q2W) from baseline (day 1) through week 10 during the double-blind treatment period
  Starting at week 12, and continuing through week 22, participants will receive open-label alirocumab SC Q2W
  Interventions: Drug: Alirocumab
- Placebo SC Q2W (Experimental): Matching placebo SC Q2W from baseline through week 10 during the double-blind treatment period
  Starting at week 12, and continuing through week 22, participants will receive open-label alirocumab SC Q2W
  Interventions: Drug: Alirocumab; Drug: Placebo

INTERVENTIONS:
Drug: Alirocumab — Alirocumab SC Q2W
  Other Names: PRALUENT®; REGN727; SAR236553
Drug: Placebo — Matching placebo SC Q2W
  Arms: Placebo SC Q2W

SUMMARY:
The primary objective of the study is to demonstrate the reduction of low-density lipoprotein cholesterol (LDL-C) with alirocumab subcutaneous (SC) every 2 weeks (Q2W) in comparison to placebo after 12 weeks of treatment.

The secondary objectives of the study are:

* To evaluate the effect of alirocumab Q2W on other lipid parameters (ie, apolipoprotein [Apo] A-1 and B, non-high-density lipoprotein cholesterol [non-HDL-C], total-cholesterol [TC], proportion of participants with 15%, 30%, and 50% LDL-C reductions, Lp(a), HDL-C, triglycerides [TG]) in participants with HoFH
* To evaluate the safety and tolerability of alirocumab SC Q2W in participants with HoFH
* To assess the pharmacokinetics of alirocumab SC Q2W in participants with HoFH
* To assess the potential development of anti-drug (alirocumab) antibodies

ELIGIBILITY:
Note: The information listed below is not intended to contain all considerations relevant to a patient's potential participation in this clinical trial, therefore not all inclusion/exclusion criteria are listed.

Key Inclusion Criteria

1. Diagnosis of HoFH by at least 1 of the following genotype or clinical criteria (all patients on LDL apheresis must be diagnosed based on genotype):

   1. Documented homozygous or compound heterozygous mutations in both low-density lipoprotein receptor (LDLR) alleles
   2. Presence of homozygous or compound heterozygous mutations in Apo B, PCSK9 or LDL receptor adaptor protein 1 (LDLRAP1)
   3. Presence of double heterozygous mutations, i.e, mutations on different genes in the LDLR, Apo B or PCSK9 alleles
   4. Untreated TC >500 mg/dL (12.93 mmol/L) and TG <300 mg/dL (3.39 mmol/L) AND Both parents with history of TC >250 mg/dL (6.46 mmol/L) OR cutaneous or tendinous xanthoma before age 10
2. Receiving a stable dose of a statin at the screening visit (documentation if statin ineffective or patient unable to tolerate statin)
3. If undergoing LDL apheresis, must have initiated LDL apheresis at least 3 months prior to screening and must have been on a stable weekly (every 7 days) or every other week (every 14 days) schedule or stable settings for at least 8 weeks

Key Exclusion Criteria:

1. Documented evidence of a null mutation in both LDLR alleles
2. Use of a PCSK9 inhibitor within 10 weeks from screening visit
3. Background medical lipid modifying therapy (LMT) that has not been stable for at least 4 weeks (6 weeks for fibrates, 24 weeks for mipomersen, 12 weeks for maximum tolerated dose of lomitapide) before the screening visit.
4. LDL apheresis schedule/apheresis settings that have not been stable for at least 8 weeks before the screening visit or an apheresis schedule/settings that is not anticipated to be stable over the next 24 weeks.
5. Use of nutraceuticals or over-the-counter (OTC) therapies known to affect lipids, at a dose/amount that has not been stable for at least 4 weeks prior to the screening visit or between the screening and randomization visits.
6. Chronic use of systemic corticosteroids, unless on a stable regimen of 10 mg daily prednisone equivalent or less for at least 6 weeks prior to randomization. Note: topical, intra-articular, nasal, inhaled and ophthalmic steroid therapies are not considered as 'systemic' and are allowed
7. Systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg at the screening visit (1 repeat measurement is allowed).
8. LDL-C level <70 mg/dL (1.81 mmol/L) at the screening visit
9. History of a myocardial infarction (MI), unstable angina leading to hospitalization, coronary artery bypass graft surgery, percutaneous coronary intervention , uncontrolled cardiac arrhythmia, carotid surgery or stenting, stroke, transient ischemic attack, valve replacement surgery, carotid revascularization, endovascular procedure or surgical intervention for peripheral vascular disease within 3 months prior to the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2020-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (26):
- United States (4):
  - Regeneron Research Site, Boca Raton, Florida
  - Regeneron Research Site, New York, New York
  - Regeneron Research Site, Cincinnati, Ohio
  - Regeneron Study Site, Dallas, Texas
- Regeneron Research Site, Innsbruck, Tyrol, Austria
- Canada (2):
  - Regeneron Research Site, Chicoutimi, Quebec
  - Regeneron Research Site, Québec, Quebec
- Regeneron Research Site, Prague, Czechia
- France (2):
  - Regeneron Research Site, Marseille
  - Regeneron Research Site, Paris
- Regeneron Research Site, Berlin, Germany
- Greece (2):
  - Regeneron Research Site, Athens
  - Regeneron Research Site, Ioannina
- Italy (2):
  - Regeneron Research Site, Napoli
  - Regeneron Research Site, Roma
- Japan (3):
  - Regeneron Research Site, Nishinomiya, Hyōgo
  - Regeneron Research Site, Kanazawa, Ishikawa-ken
  - Regeneron Research Site, Suita, Osaka
- South Africa (2):
  - Regeneron Research Site, Parktown, Johannesburg
  - Regeneron Research Site, Cape Town, Western Cape
- Regeneron Study Site, Taipei, Taiwan
- Turkey (Türkiye) (2):
  - Regeneron Research Site, Beşevler, Ankara
  - Regeneron Research Site, Izmir, Bornova
- Ukraine (3):
  - Regeneron Research Site, Ivano-Frankivsk
  - Regeneron Research Site, Kharkiv
  - Regeneron Research Site, Kyiv

REFERENCES:
- [Derived] Blom DJ, Harada-Shiba M, Rubba P, Gaudet D, Kastelein JJP, Charng MJ, Pordy R, Donahue S, Ali S, Dong Y, Khilla N, Banerjee P, Baccara-Dinet M, Rosenson RS. Efficacy and Safety of Alirocumab in Adults With Homozygous Familial Hypercholesterolemia: The ODYSSEY HoFH Trial. J Am Coll Cardiol. 2020 Jul 14;76(2):131-142. doi: 10.1016/j.jacc.2020.05.027. PMID 32646561

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 27 centers in 13 countries around Europe, Asia, South Africa, and North America. A total of 85 participants were screened. Of those,16 were considered screen failures (mainly due to violations of inclusion/exclusion criteria).
Pre-assignment Details: Sixty-nine of the 85 participants were eligible and randomized in a 2:1 ratio to receive either alirocumab 150 mg SC Q2W or matching placebo. Randomization was stratified by LDL apheresis treatment status (on vs off treatment).
Groups:
- Placebo in DBTP: Participants received matching placebo subcutaneously (SC) every 2 weeks (Q2W) from baseline (Day 1) through Week 10 during the double-blind treatment period. Starting at Week 12, and continuing through Week 22, all participants received open-label alirocumab SC Q2W
- Alirocumab 150 mg SC Q2W: Participants in this arm received alirocumab 150 milligrams (mg) SC Q2W from baseline (Day 1) through Week 10 during the double-blind treatment period. Starting at Week 12, and continuing through Week 22, all participants received open-label alirocumab SC Q2W
Period: Double-Blind Treatment Period (DBTP)
Arm/Group | Placebo in DBTP | Alirocumab 150 mg SC Q2W
Started | 24 | 45
Completed | 24 | 45
Not Completed | 0 | 0
Period: Open-Label Treatment Period (OLTP)
Arm/Group | Placebo in DBTP | Alirocumab 150 mg SC Q2W
Started | 24 | 45
Completed | 24 | 42
Not Completed | 0 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo in DBTP | Alirocumab 150 mg SC Q2W | Total
Number analyzed (Participants) | 24 | 45 | 69
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.4 (15.80) | 42.3 (14.13) | 43.4 (14.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 24 | 35
  Male | 13 | 21 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 24 | 43 | 67
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 18 | 36 | 54
  Black or African American | 0 | 2 | 2
  Asian | 5 | 7 | 12
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 1 | 0 | 1
Low-density lipoprotein cholesterol (LDL-C) [Mean (Standard Deviation); unit: milligram/deciLiter (mg/dL)] | 259.6 (175.75) | 295.0 (154.59) | 282.7 (161.86)
Non-high-density lipoprotein cholesterol (Non-HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 282.0 (177.41) | 320.5 (160.36) | 307.1 (166.22)
Total-cholesterol (Total-C) [Mean (Standard Deviation); unit: mg/dL] | 325.1 (171.57) | 364.3 (157.30) | 350.7 (162.24)
High-density lipoprotein cholesterol (HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 43.2 (11.96) | 43.8 (14.78) | 43.6 (13.78)
Fasting triglycerides (TG) [Mean (Standard Deviation); unit: mg/dL] | 111.7 (77.97) | 128.0 (74.34) | 122.3 (75.45)
Lipoprotein(a) [Lp(a)] [Mean (Standard Deviation); unit: mg/dL] | 40.0 (36.41) | 42.9 (36.34) | 41.9 (36.12)
Apolipoprotein-B (Apo-B) [Mean (Standard Deviation); unit: mg/dL] | 175.0 (95.12) | 193.3 (87.59) | 186.9 (90.01)
Apolipoprotein-A1 (Apo-A1) [Mean (Standard Deviation); unit: mg/dL] | 124.8 (24.59) | 125.6 (28.57) | 125.3 (27.07)
Apo-B/Apo-A1 [Mean (Standard Deviation); unit: ratio] | 1.590 (1.4746) | 1.635 (0.8693) | 1.619 (1.1067)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Low-density Lipoprotein Cholesterol (LDL-C) From Baseline to Week 12 (Intent-to-Treat [ITT] Estimand)
Description: The percent change in LDL-C from baseline to week 12 is defined as: 100x (LDL-C value at week 12 - LDL-C value at baseline) / LDL-C value at baseline.
Time Frame: Baseline to Week 12
Population: ITT estimand (All randomized participants who had at least 1 measurement value for LDL-C before the first dose of double blind investigational study drug)
Measure: Least Squares Mean (Standard Error); unit: Percentage of change
Arm/Group | Placebo in DBTP | Alirocumab 150 mg SC Q2W
Number analyzed (Participants) | 24 | 45
Percentage of change | 8.6 (6.3) | -26.9 (4.6)
Statistical Analysis 1: Comparison: Placebo in DBTP vs Alirocumab 150 mg SC Q2W; Test type: Superiority; p < 0.0001, MMRM — P-value taken from MMRM (mixed-effect model with repeated measures) analysis; Least squares (LS) mean difference = -35.6, 95% CI 2-sided [-51.2 to -19.9], Standard Error of Mean 7.8 — p-value vs Placebo

2. Secondary Outcome: Percent Change in Apolipoprotein (Apo) B From Baseline to Week 12 (ITT Estimand)
Description: ITT estimand; The percent change in Apo B from baseline to week 12 is defined as: 100x (Apo B value at week 12 - Apo B value at baseline) / Apo B value at baseline.
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: Percentage of change
Arm/Group | Placebo in DBTP | Alirocumab 150 mg SC Q2W
Number analyzed (Participants) | 24 | 45
Percentage of change | 7.2 (5.0) | -22.5 (3.7)
Statistical Analysis 1: Comparison: Placebo in DBTP vs Alirocumab 150 mg SC Q2W; Test type: Superiority; p < 0.0001, MMRM — p-value taken from MMRM (mixed-effect model with repeated measures) analysis; Least squares (LS) mean difference = -29.8, 95% CI 2-sided [-42.3 to -17.3], Standard Error of Mean 6.3

3. Secondary Outcome: Percent Change in Non-high-density Lipoprotein Cholesterol (Non-HDL-C) From Baseline to Week 12
Description: ITT estimand; The percent change in non-HDL-C from baseline to week 12 is defined as: 100x (non-HDL-C value at week 12 - non-HDL-C value at baseline) / non-HDL-C value at baseline.
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: Percentage of change
Arm/Group | Placebo in DBTP | Alirocumab 150 mg SC Q2W
Number analyzed (Participants) | 24 | 45
Percentage of change | 8.0 (5.9) | -24.8 (4.3)
Statistical Analysis 1: Comparison: Placebo in DBTP vs Alirocumab 150 mg SC Q2W; Test type: Superiority; p < 0.0001, MMRM — P-value taken from MMRM (mixed-effect model with repeated measures) analysis; Least squares (LS) mean difference = -32.9, 95% CI 2-sided [-47.6 to -18.2], Standard Error of Mean 7.4

4. Secondary Outcome: Percent Change in Total Cholesterol (TC) From Baseline to Week 12
Description: ITT estimand; The percent change in TC from baseline to week 12 is defined as: 100x (TC value at week 12 - TC value at baseline) / TC value at baseline.
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: Percentage of change
Arm/Group | Placebo in DBTP | Alirocumab 150 mg SC Q2W
Number analyzed (Participants) | 24 | 45
Percentage of change | 6.6 (5.0) | -19.8 (3.7)
Statistical Analysis 1: Comparison: Placebo in DBTP vs Alirocumab 150 mg SC Q2W; Test type: Superiority; p < 0.0001, MMRM — P-value taken from MMRM (mixed-effect model with repeated measures) analysis; Least squares (LS) mean difference = -26.5, 95% CI 2-sided [-38.9 to -14.0], Standard Deviation 6.2

5. Secondary Outcome: Percentage of Participants With ≥15% Reduction in LDL-C at Week 12
Description: ITT estimand
Time Frame: At Week 12
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo in DBTP | Alirocumab 150 mg SC Q2W
Number analyzed (Participants) | 24 | 45
Percentage of participants | 12.5 | 61.9
Statistical Analysis 1: Comparison: Placebo in DBTP vs Alirocumab 150 mg SC Q2W; Test type: Superiority; p = 0.0004, Regression, Logistic; Odds Ratio, log = 12.2, 95% CI 2-sided [3.1 to 48.8]

6. Secondary Outcome: Percentage of Participants With ≥30% Reduction in LDL-C at Week 12
Description: ITT estimand
Time Frame: At Week 12
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo in DBTP | Alirocumab 150 mg SC Q2W
Number analyzed (Participants) | 24 | 45
Percentage of participants | 4.2 | 57.1
Statistical Analysis 1: Comparison: Placebo in DBTP vs Alirocumab 150 mg SC Q2W; Test type: Superiority; p = 0.0010, Regression, Logistic; Odds Ratio, log = 36.5, 95% CI 2-sided [4.3 to 308.9]

7. Secondary Outcome: Percent Change in Lipoprotein(a) [Lp(a)] From Baseline to Week 12
Description: ITT estimand; The percent change in Lp(a) from baseline to week 12 is defined as: 100x (Lp(a) value at week 12 - Lp(a) value at baseline) / Lp(a) value at baseline.
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: Percentage of change
Arm/Group | Placebo in DBTP | Alirocumab 150 mg SC Q2W
Number analyzed (Participants) | 24 | 45
Percentage of change | 8.8 (5.4) | -19.6 (4.0)
Statistical Analysis 1: Comparison: Placebo in DBTP vs Alirocumab 150 mg SC Q2W; Test type: Superiority; p < 0.0001, Regression model; Mean Difference (Final Values) = -28.4, 95% CI 2-sided [-41.5 to -15.2], Standard Deviation 6.7

8. Secondary Outcome: Percentage of Participants With ≥50% Reduction in LDL-C at Week 12
Description: ITT estimand
Time Frame: At Week 12
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo in DBTP | Alirocumab 150 mg SC Q2W
Number analyzed (Participants) | 24 | 45
Percentage of participants | 0 | 26.7
Statistical Analysis 1: Comparison: Placebo in DBTP vs Alirocumab 150 mg SC Q2W; Test type: Superiority; p = 0.0017, Exact Conditional Logistic Regression; Odds Ratio (OR) = 17.7, 95% CI 2-sided [lower limit 3.3] (Maximum likelihood estimate does not exist)

9. Secondary Outcome: Percent Change in HDL-C From Baseline to Week 12 - ITT Analysis
Description: ITT estimand; The percent change in HDL-C from baseline to week 12 is defined as: 100x (HDL-C value at week 12 - HDL-C value at baseline) / HDL-C value at baseline.
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: Percentage of change
Arm/Group | Placebo in DBTP | Alirocumab 150 mg SC Q2W
Number analyzed (Participants) | 24 | 45
Percentage of change | 2.7 (3.1) | 6.3 (2.3)
Statistical Analysis 1: Comparison: Placebo in DBTP vs Alirocumab 150 mg SC Q2W; Test type: Superiority; p = 0.3541, MMRM — P-value taken from MMRM (mixed-effect model with repeated measures) analysis; Least squares (LS) mean difference = 3.6, 95% CI 2-sided [-4.1 to 11.3], Standard Error of Mean 3.8

10. Secondary Outcome: Percent Change in Fasting Triglycerides (TG) From Baseline to Week 12
Description: ITT estimand; The percent change in TG from baseline to week 12 is defined as: 100x (TG value at week 12 - TG value at baseline) / TG value at baseline.
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: Percentage of change
Arm/Group | Placebo in DBTP | Alirocumab 150 mg SC Q2W
Number analyzed (Participants) | 24 | 45
Percentage of change | 3.9 (5.7) | -7.4 (4.2)
Statistical Analysis 1: Comparison: Placebo in DBTP vs Alirocumab 150 mg SC Q2W; Test type: Superiority; Mean Difference (Final Values) = -11.3, 95% CI 2-sided [-25.2 to 2.6], Standard Error of Mean 7.1

11. Secondary Outcome: Percent Change in Apo A-1 From Baseline to Week 12 -- ITT Analysis
Description: ITT estimand; The percent change in Apo A-1 from baseline to week 12 is defined as: 100x (Apo A-1 value at week 12 - Apo A-1 value at baseline) / Apo A-1 value at baseline.
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: Percentage of change
Arm/Group | Placebo in DBTP | Alirocumab 150 mg SC Q2W
Number analyzed (Participants) | 24 | 45
Percentage of change | 1.4 (2.9) | 5.0 (2.1)
Statistical Analysis 1: Comparison: Placebo in DBTP vs Alirocumab 150 mg SC Q2W; Test type: Superiority; Least squares (LS) mean difference = 3.6, 95% CI 2-sided [-3.6 to 10.7], Standard Deviation 3.6

12. Secondary Outcome: Percent Change in LDL-C From Baseline to Week 12 (On-treatment Estimand)
Description: Percent change for LDL-C from baseline to Week 12 during the efficacy treatment period, which is defined as the time from the first double-blind investigational study drug injection up to 21 days after the last double-blind investigational study drug injection, or the first dose of the open-label investigational study drug, whichever is earlier.
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: Percentage of change
Arm/Group | Placebo in DBTP | Alirocumab 150 mg SC Q2W
Number analyzed (Participants) | 24 | 45
Percentage of change | 8.6 (6.3) | -26.9 (4.6)
Statistical Analysis 1: Comparison: Placebo in DBTP vs Alirocumab 150 mg SC Q2W; Test type: Superiority; Least squares (LS) mean difference = -35.6, 95% CI 2-sided [-51.2 to -19.9], Standard Error of Mean 7.8

13. Secondary Outcome: Percent Change in Apo B From Baseline to Week 12 (On-treatment Estimand)
Description: Percent change for Apo B from baseline to Week 12 during the efficacy treatment period, which is defined as the time from the first double-blind investigational study drug injection up to 21 days after the last double-blind investigational study drug injection, or the first dose of the open-label nvestigational study drug, whichever is earlier.
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: Percentage of change
Arm/Group | Placebo in DBTP | Alirocumab 150 mg SC Q2W
Number analyzed (Participants) | 24 | 45
Percentage of change | 7.2 (5.0) | -22.5 (3.7)
Statistical Analysis 1: Comparison: Placebo in DBTP vs Alirocumab 150 mg SC Q2W; Test type: Superiority; Least squares (LS) mean difference = -29.8, 95% CI 2-sided [-43.3 to -17.3], Standard Error of Mean 6.3

14. Secondary Outcome: Percent Change in Non-HDL-C From Baseline to Week 12 (On-treatment Estimand)
Description: Percent change for non-HDL-C from baseline to Week 12 during the efficacy treatment period, which is defined as the time from the first double-blind investigational study drug injection up to 21 days after the last double-blind investigational study drug injection, or the first dose of the open-label investigational study drug, whichever is earlier.
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: Percentage of change
Arm/Group | Placebo in DBTP | Alirocumab 150 mg SC Q2W
Number analyzed (Participants) | 24 | 45
Percentage of change | 8.0 (5.9) | -24.8 (4.3)
Statistical Analysis 1: Comparison: Placebo in DBTP vs Alirocumab 150 mg SC Q2W; Test type: Superiority; Least squares (LS) mean difference = -32.9, 95% CI 2-sided [-47.6 to -18.2], Standard Error of Mean 7.4

15. Secondary Outcome: Percent Change in TC From Baseline to Week 12 (On-treatment Estimand)
Description: Percent change for TC from baseline to Week 12 during the efficacy treatment period, which is defined as the time from the first double-blind investigational study drug injection up to 21 days after the last double-blind investigational study drug injection, or the first dose of the open-label investigational study drug, whichever is earlier.
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: Percentage of change
Arm/Group | Placebo in DBTP | Alirocumab 150 mg SC Q2W
Number analyzed (Participants) | 24 | 45
Percentage of change | 6.6 (5.0) | -19.8 (3.7)
Statistical Analysis 1: Comparison: Placebo in DBTP vs Alirocumab 150 mg SC Q2W; Test type: Superiority; Least squares (LS) mean difference = -26.5, 95% CI 2-sided [-28.9 to -14.0], Standard Error of Mean 6.2

16. Secondary Outcome: Percent Change in Lp(a) From Baseline to Week 12 (On-treatment Estimand)
Description: Percent change for LP(a) from baseline to Week 12 during the efficacy treatment period, which is defined as the time from the first double-blind investigational study drug injection up to 21 days after the last double-blind investigational study drug injection, or the first dose of the open-label investigational study drug, whichever is earlier.
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: Percentage of change
Arm/Group | Placebo in DBTP | Alirocumab 150 mg SC Q2W
Number analyzed (Participants) | 24 | 45
Percentage of change | 8.8 (5.4) | -19.6 (4.0)
Statistical Analysis 1: Comparison: Placebo in DBTP vs Alirocumab 150 mg SC Q2W; Test type: Superiority; Mean Difference (Final Values) = -28.4, 95% CI 2-sided [-41.5 to -15.2], Standard Error of Mean 6.7

17. Secondary Outcome: Percent Change in HDL-C From Baseline to Week 12 (On-treatment Estimand)
Description: Percent change for HDL-C from baseline to Week 12 during the efficacy treatment period, which is defined as the time from the first double-blind investigational study drug injection up to 21 days after the last double-blind investigational study drug injection, or the first dose of the open-label investigational study drug, whichever is earlier.
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: Percentage of change
Arm/Group | Placebo in DBTP | Alirocumab 150 mg SC Q2W
Number analyzed (Participants) | 24 | 45
Percentage of change | 2.7 (3.1) | 6.3 (2.3)
Statistical Analysis 1: Comparison: Placebo in DBTP vs Alirocumab 150 mg SC Q2W; Test type: Superiority; Least squares (LS) mean difference = 3.6, 95% CI 2-sided [-4.1 to 11.3], Standard Error of Mean 3.8

18. Secondary Outcome: Percent Change in Fasting TG From Baseline to Week 12 (On-treatment Estimand)
Description: Percent change for fasting TG from baseline to Week 12 during the efficacy treatment period, which is defined as the time from the first double-blind investigational study drug injection up to 21 days after the last double-blind investigational study drug injection, or the first dose of the open-label investigational study drug, whichever is earlier.
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: Percentage of change
Arm/Group | Placebo in DBTP | Alirocumab 150 mg SC Q2W
Number analyzed (Participants) | 24 | 45
Percentage of change | 3.9 (5.7) | -7.4 (4.2)
Statistical Analysis 1: Comparison: Placebo in DBTP vs Alirocumab 150 mg SC Q2W; Test type: Superiority; Mean Difference (Final Values) = -11.3, 95% CI 2-sided [-25.2 to 2.6], Standard Error of Mean 7.1

19. Secondary Outcome: Percent Change in Apo A-1 From Baseline to Week 12 (On-treatment Estimand)
Description: Percent change for Apo A-1 from baseline to Week 12 during the efficacy treatment period, which is defined as the time from the first double-blind investigational study drug injection up to 21 days after the last double-blind investigational study drug injection, or the first dose of the open-label investigational study drug, whichever is earlier.
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: Percentage of change
Arm/Group | Placebo in DBTP | Alirocumab 150 mg SC Q2W
Number analyzed (Participants) | 24 | 45
Percentage of change | 1.4 (2.9) | 5.0 (2.1)
Statistical Analysis 1: Comparison: Placebo in DBTP vs Alirocumab 150 mg SC Q2W; Test type: Superiority; Least squares (LS) mean difference = 3.6, 95% CI 2-sided [-3.6 to 10.7], Standard Error of Mean 3.6

20. Secondary Outcome: Percentage of Participants With ≥15% Reduction, ≥30% Reduction, and ≥50% Reduction in LDL-C at Week 12 (On-treatment Estimand)
Time Frame: At Week 12
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo in DBTP | Alirocumab 150 mg SC Q2W
Number analyzed (Participants) | 24 | 45
Percentage of participants
  ≥ 15% | 12.5 | 61.9
  ≥ 30% | 4.2 | 57.1
  ≥ 50% | 0 | 26.7
Statistical Analysis 1: Comparison: Placebo in DBTP vs Alirocumab 150 mg SC Q2W; ≥15% reduction; Test type: Superiority; Odds Ratio (OR) = 12.2, 95% CI 2-sided [3.1 to 48.8]
Statistical Analysis 2: Comparison: Placebo in DBTP vs Alirocumab 150 mg SC Q2W; Test type: Superiority — ≥ 30% reduction; Odds Ratio (OR) = 36.5, 95% CI 2-sided [4.3 to 308.9]
Statistical Analysis 3: Comparison: Placebo in DBTP vs Alirocumab 150 mg SC Q2W; ≥ 50% reduction; Test type: Superiority; Odds Ratio (OR) = 17.7, 95% CI 2-sided [lower limit 3.3] (Maximum likelihood estimate does not exist)

21. Secondary Outcome: Absolute Change in the Ratio of Apo B/Apo A-1 From Baseline to Week 12 (ITT Estimand)
Description: Ratio of Apo B/Apo A1 at week 12 minus ratio of Apo B/Apo A1 at baseline
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: Ratio of change
Arm/Group | Placebo in DBTP | Alirocumab 150 mg SC Q2W
Number analyzed (Participants) | 24 | 45
Ratio of change | 0.0 (0.1) | -0.3 (0.1)
Statistical Analysis 1: Comparison: Placebo in DBTP vs Alirocumab 150 mg SC Q2W; Test type: Superiority; Least squares (LS) mean difference = -0.3, 95% CI 2-sided [-0.6 to -0.1], Standard Error of Mean 0.1

22. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADA) to REGN727 Over Time
Time Frame: 26 weeks
Population: Here 'n' = number of evaluable participants at this time point
Measure: Number; unit: Participants
Arm/Group | Placebo in DBTP | Alirocumab 150 mg SC Q2W
Number analyzed (Participants) | 24 | 44
Participants | 1 | 1

23. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: All AEs will be recorded from time of informed consent to end of study. Only treatment-emergent adverse events (TEAE) will be reported. Double-blind TEAE observation period is defined as time from first dose of double-blind study drug to last dose of double-blind study drug +70 days, or up to day before first dose of open-label study drug administration, whichever is earlier. Open-label TEAE observation period is defined as time from first open-label study treatment administration to last open-label study treatment administration +70 days.
Time Frame: Baseline to week 32 (End of Study)
Measure: Number; unit: Participants
Groups:
- Alirocumab 150 mg SC Q2W in OLTP: Participants who received at least 1 dose or part of a dose of open-label investigational study drug alirocumab in OLTP
Arm/Group | Placebo in DBTP | Alirocumab 150 mg SC Q2W | Alirocumab 150 mg SC Q2W in OLTP
Number analyzed (Participants) | 24 | 45 | 69
Participants
  Participants with any TEAE | 12 | 20 | 24
  Participants with TEAE Serious Adverse Event (SAE) | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) to end of study (Day 225)
Groups:
- DB Placebo (DBTP): Participants received matching placebo subcutaneously (SC) every 2 weeks (Q2W) from baseline (Day 1) through Week 10 during the double-blind treatment period.
- DB Alirocumab 150 Q2W (DBTP): Participants in this arm received alirocumab 150 milligrams (mg) SC Q2W from baseline (Day 1) through Week 10 during the double-blind treatment period.
- DB Placebo (OLTP): Participants received matching placebo subcutaneously (SC) every 2 weeks (Q2W) from baseline (Day 1) through Week 10 during the double-blind treatment period. Starting at Week 12, and continuing through Week 22, all participants received open-label alirocumab SC Q2W
- DB Alirocumab 150 Q2W (OLTP): Participants in this arm received alirocumab 150 milligrams (mg) SC Q2W from baseline (Day 1) through Week 10 during the double-blind treatment period. Starting at Week 12, and continuing through Week 22, all participants received open-label alirocumab SC Q2W
Arm/Group | DB Placebo (DBTP) | DB Alirocumab 150 Q2W (DBTP) | DB Placebo (OLTP) | DB Alirocumab 150 Q2W (OLTP)
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/45 | 0/24 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/45 | 0/24 | 1/45
Other Adverse Events (participants affected / at risk) | 4/24 | 8/45 | 2/24 | 4/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB Placebo (DBTP) (N=24) | DB Alirocumab 150 Q2W (DBTP) (N=45) | DB Placebo (OLTP) (N=24) | DB Alirocumab 150 Q2W (OLTP) (N=45)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB Placebo (DBTP) (N=24) | DB Alirocumab 150 Q2W (DBTP) (N=45) | DB Placebo (OLTP) (N=24) | DB Alirocumab 150 Q2W (OLTP) (N=45)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (3) | 1 (1) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (8) | 2 (2) | 1 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2019-01-04): https://cdn.clinicaltrials.gov/large-docs/21/NCT03156621/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/21/NCT03156621/SAP_001.pdf